CLINICAL TRIAL: NCT06489236
Title: Effectiveness of an Intervention on Vaccine Hesitancy Among Pediatric Nurses and Pediatricians: A Mixed Methods Study
Brief Title: Effectiveness of an Intervention on Vaccine Hesitancy Among Pediatric Nurses and Pediatricians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Public Health Agency of Barcelona (Other); Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Elia Diez David, Principal Investigator, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI21/01710
Record Dates: First submitted 2024-06-14; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Vaccination Hesitancy; Pediatric ALL; Presumptive Communication; Motivational Interviewing
MeSH Terms: conditions — Vaccination Hesitancy; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Public primary care center pediatric teams in Barcelona city and Central Catalonia that enroll in the study will be randomly allocated into two parallel groups: intervention and control groups. This allocation will be conducted through a web-based procedure by block design. Pediatric teams will be paired based on the assigned population under 14 years old, the socioeconomic status of the basic health area, immunization coverage, and location, using data from the Primary Care Services Information System (SISAP). Team names will be blinded throughout the randomization process. Once randomization is complete, allocation will be unblinded to the research team. The control group will follow the standard procedures for vaccination promotion and vaccine hesitancy management. Pediatric teams in the control group will be offered the intervention once it has been evaluated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccination promotion training program (Experimental): Pediatric nurses and pediatricians enrolled in the study employed at public primary care centers in Barcelona city and Central Catalonia randomly allocated to the intervention group. Intervention administered: 12-hour, medically accredited, evidence-based training program focused on vaccination promotion.
  Interventions: Behavioral: Vaccine Confidence: Skills to Promote Vaccination in the Pediatric Consultations
- Practice as usual (No Intervention): Pediatric nurses and pediatricians enrolled in the study employed at public primary care centers in Barcelona city and Central Catalonia randomly allocated to the control group. No intervention administered. Practice as usual.

INTERVENTIONS:
Behavioral: Vaccine Confidence: Skills to Promote Vaccination in the Pediatric Consultations — Intervention mapping principles guided a multidisciplinary team through the development of the intervention. The intervention is a 12-hour training program focused on improving vaccination promotion and vaccine hesitancy management during pediatric consultations. The program comprises 10 hours of online education and 2 hours of in-person activities. Online training materials (short video lectures, video case studies, and readings) were structured in three learning modules covering vaccine and vaccine hesitancy technical information, vaccination promotion communication strategies, and practice organizational resources. In-person activities involved role-playings and group discussions. Intervention content is evidence-based. As a participation incentive, pediatric nurses and pediatricians who complete all program activities, including a multiple-choice final test, will receive 2,5 accredited continuing medical education credits.
  Arms: Vaccination promotion training program

SUMMARY:
The objective of this cluster randomized controlled trial is to assess the effectiveness of a multicomponent intervention designed to improve pediatric nurses' and pediatricians' knowledge, self-efficacy, communication skills, and practice administrative procedures and policies for promoting vaccines in the child and adolescent immunization schedule and addressing patient vaccine hesitancy.

The main research questions are:

* Does the intervention meet pediatric nurses' and pediatricians' educational needs regarding vaccination?
* Does the intervention increase the use of presumptive communication by pediatric nurses and pediatricians during vaccine conversations?
* Does the intervention enhance the confidence of pediatric nurses and pediatricians to effectively navigate conversations with vaccine-hesitant families?
* Does the intervention enhance the abilities of pediatric nurses and pediatricians to effectively navigate conversations with vaccine-hesitant families?

Participants assigned to the intervention group will complete a 12-hour, medically accredited, evidence-based training program focused on vaccination promotion. This training will be divided into two components: 10 hours of online education covering vaccines and vaccination communication strategies, and 2 hours of in-person activities involving role-playing and group discussions. Pediatric nurses and pediatricians assigned to the control group will continue with their usual practices. To assess the effectiveness of the intervention formative and pre/post summative evaluations with a mixed-methods approach will be carried out.

DETAILED DESCRIPTION:
Background/Objectives/Hypothesis:

How pediatric nurses and pediatricians (PN&P) handle vaccination conversations can significantly influence vaccination decisions. PN&P, who are at the frontline of administering childhood vaccinations, may not be well-equipped to address vaccination doubts or concerns of parents or legal guardians. A study conducted among PN&P in primary care centers in Barcelona revealed that only 71% of professionals, felt they had sufficient training, information, and resources to adequately respond to questions from vaccine-hesitant families. This lack of preparedness was reported by 40% of nurses and 17% of pediatricians. Additionally, PN&P also expressed a need for more information about vaccines in online (52.3%) or through in-person training sessions (50.2%).

Intervention mapping (IM) is a theory- and evidenced-based iterative tool useful in the planning of health promotion interventions. Using the IM framework, the investigators developed a 12-hour training program to increase PN&P's knowledge, self-efficacy, communication skills and organizational culture for improving vaccination promotion and vaccine hesitancy management during pediatric consultations. The program comprises 10 hours of online education and 2 hours of in-person activities. Online training materials include short video lectures, video case studies, and readings. In-person activities involve role-playings and group discussions. The program was accredited by the Catalan Council for Continuing Education of Health Professions (CCFCPS). To incentivize participation, providers completing all program activities, including a multiple-choice final test, will receive 2.5 accredited continuing medical education credits.

Mixed-methods evaluations provide a more comprehensive and profound understanding of intervention effects and help identify areas for improvement. This study aims to evaluate the effectiveness of an intervention on PN&P psychosocial determinants (knowledge, beliefs, attitudes, and self-efficacy) and behaviors in promoting vaccination and addressing vaccine hesitancy during pediatric consultations using quantitative and qualitative methods. Specifically, the investigators will assess PN&P's satisfaction with the 12-hour training program and changes in their psychosocial determinants and vaccination behaviors.

Methods:

The investigators will employ a mixed-method approach for the evaluation of the intervention. Quantitative and qualitative data will be integrated through triangulation principles. Quantitative analysis will involve the design of a two-arm cluster randomized control trial. For the qualitative evaluation, the investigators plan to carry out a descriptive qualitative study with a phenomenological approach.

Cluster Randomized Control Trial

Study design: Two-arm parallel cluster randomized controlled trial during 5 months with pediatric care providers in public primary care centers in Barcelona city (Catalonia, Spain) and Central Catalonia (Catalonia, Spain). Intervention group will receive a 12-hour online and in-person training program for improving vaccination promotion and vaccine hesitancy management during pediatric consultations.

Randomization: Pediatric teams will be paired based on the assigned population under 14 years old, the socioeconomic status of the basic health area, immunization coverage, and location using data from the Primary Care Services Information System (SISAP). Randomization will be carried out with a block design. Team names will be blinded throughout the randomization process. Once randomization is complete, allocation will be unblinded to the research team. The control group will follow the standard procedures for vaccination promotion and vaccine hesitancy management.

Population and sample: Pediatric nurses and pediatricians (PN&P) involved in the administration of systematic childhood vaccines and working in primary care centers in Barcelona city (N= 41 centers, N= 342 pediatric care providers) and Central Catalonia (N=38 centers, N= 108 pediatric care providers). For the recruitment, the research team will contact the Head of Pediatrics in each of the regions where the training is planned to be implemented. Study participation will be offered after agreement of the primary care centers. An information session will be held to ensure participants understand the study's purposes, procedures, and timeline, as well as to address questions or potential concerns. Based on previous research conducted with PN&P in Barcelona, the investigators estimate a baseline self-efficacy related to vaccination promotion and vaccine-hesitant management of 71%. The investigators assume this percentage to be similar for PN&P in Central Catalonia. Accepting an alpha risk of 0.05 and a beta risk of 0.2 in a bilateral contrast, 82 subjects in each group will be able to detect a statistically significant difference of 18% with an estimated loss of follow-up rate of 10%. Since randomization will be done by clusters, a cluster effect of 1.65 will be applied to the sample size, resulting in an overall sample of 270 participants (135 per group). Therefore, the study will be powered enough to detect at least a difference of 18% in PN&P's self-efficacy.

Recruitment: PN&P will enlist in the study by completing a brief online form available via Microsoft Forms. This form will be accessible through the study's information brochure and shared in the online information session. Upon receiving the applications, the research team will grant participants access to the online learning platform (Moodle). To complete the enrollment, all participants will have to read the participant information sheet and provide signed informed consent.

Data collection: PN&P will be asked to complete a baseline and post-intervention questionnaire available on the online learning platform after enrollment and intervention periods. The questionnaire has been built based on previously validated scales from existing literature and has been pre-tested and piloted. As the questionnaires will be self-administered, the research team will perform daily checks to ensure data quality and completeness. The questionnaires will collect PN&P's knowledge on vaccine safety and effectiveness, key childhood immunization beliefs, self-efficacy in managing vaccine-hesitant situations, frequency of vaccine promotion behaviors during pediatric consultations, practice immunization organization culture, as well as standard demographic information (age, sex, professional role, years of practice, offspring, and region). PN&P's psychosocial determinants and vaccination promotion behaviors will be measured using five-point Likert scales. Data will be securely handled and stored to maintain confidentiality, with access restricted to the research team members only.

Statistical analysis plan: Analyses will be performed by intention to treat, including all subjects in the randomized pediatric teams, and per protocol. Differences between pre-post measures within intervention and control groups will be assessed with multivariate logistic regression models. Models will be adjusted by baseline values, age, sex, having offspring, profession, and years of professional practice. Statistical significance will be set at α<0.05. Analysis will be performed using R software (version 4.3.0).

Qualitative study

Study design: Descriptive qualitative study with a phenomenological design approach.

Population and sample: PN&P in public primary care centers in Barcelona city (Catalonia, Spain) and Central Catalonia (Catalonia, Spain). Sampling units will be chosen based on theoretically predefined profiles. In this study, the professional role in pediatric care (medicine or nursing) may influence experiences and discourse regarding intervention satisfaction and outcomes. To prevent professional hierarchy from interfering, the groups will be segmented by type of professional (nurses and pediatricians). The investigators will use criterion sampling to select PN&P who have successfully completed the training program. Participants will be selected considering discursive heterogeneity based on criteria including gender, years of professional experience, rurality, offspring, socioeconomic status of the basic health area, number of attempts to pass the program's exam, and overall degree of satisfaction with the training program. To achieve data saturation, the investigators plan to conduct four discussion groups: two with pediatric nursing staff and two with pediatric medical staff. The sampling will be cumulative and sequential, and the final sample size will be determined by the saturation of the information. Recruitment will continue until information sufficiency is reached, meaning no new themes or insights emerge from the discussions.

Recruitment: PN&P who have completed the training program will be organized into the four discussion groups based on pre-established sampling criteria. Selected individuals will receive an email invitation to participate, along with study information. Discussion groups will be scheduled to maximize participants' availability. In cases where a group does not meet the minimum required number of participants (6-8 participants per group), the research team will contact other individuals with similar profiles who meet the sampling criteria. To encourage participation, PN&P will receive a 50 euros gift card.

Data collection and management: PN&P perceptions, opinions, and experiences regarding the intervention will be explored through focus groups carried out at least three months after the conclusion of the training program. Focus groups will be held online via video calls using the Teams platform, allowing the participation of professionals from both study regions (Barcelona and Central Catalonia). Each group will be facilitated by a moderator and assisted by an observer. A semi-structured guide will ensure comprehensive exploration of all relevant topics. The topic guide will cover questions related to: (1) intervention implementation (most and least valued aspects, barriers, facilitators, satisfaction, perceived quality, and suggestions) and (2) intervention outcomes (perceived changes on communication skills, knowledge, attitudes towards vaccination, self-efficacy in consultations with vaccine-hesitant patients, and social norms). Sessions are expected to last approximately 1.5 to 2 hours and will be recorded in audio and video formats with prior verbal consent from all participants. Recordings will be securely stored, transcribed, and analyzed anonymously. Access to recordings and transcripts will be restricted to the research team.

Method of analysis: Focus groups sessions will be transcribed using the Turboscribe tool. One member of the research team will revise and verify the transcription outputs and incorporate relevant observations made by the observer into the final transcripts. The investigators will perform thematic analysis supported by ATLAS.ti software version 24.1. Analysis plan: a) identify the basic units of meaning, b) generate mixed categories based on the predefined topic guide and the emerging data, c) text coding, d) analyze content between and within categories, e) create subcategories, f) triangulate results. All stages of the coding and categorization processes will be discussed and agreed by all research team members to ensure methodological consistency and data quality.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric nurses
* Pediatricians
* Employed in public primary care centers in Barcelona city and Central Catalonia

Exclusion Criteria:

* Other health care professionals
* Not completing the study baseline questionnaire
* Changing primary care centers during the intervention period
* Not actively working for the entire duration of the intervention period (October 2023 to February 2024)

Max Age: 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Self-perceived preparedness to handle vaccination concerns during pediatric consultations | Baseline and 5 months later
  Pediatric nurses and pediatricians will complete both a baseline and post-intervention questionnaire. The outcome, "Self-perceived preparedness to handle vaccination concerns during pediatric consultations," will be evaluated using the following question: "I feel sufficiently trained to address vaccination concerns that families may raise," measured on a five-point Likert scale ranging from "strongly disagree" to "strongly agree".
Presenting vaccination as a default behavior using presumptive communication | Baseline and 5 months later
  Pediatric nurses and pediatricians will complete both a baseline and post-intervention questionnaire. The outcome, " Presenting vaccination as a default behavior using presumptive communication," will be evaluated using the following question: " I will start the vaccination conversation assuming the child will get vaccinated," measured on a five-point Likert scale ranging from "yes, always" to "never".
Explicitly recommending vaccination to vaccine hesitant families | Baseline and 5 months later
  Pediatric nurses and pediatricians will complete both a baseline and post-intervention questionnaire. The outcome, " Explicitly recommending vaccination to vaccine hesitant families," will be evaluated using the following question: " I will recommend getting vaccinated during that same visit" measured on a five-point Likert scale ranging from "yes, always" to "never".

CONTACTS AND LOCATIONS:
Overall Officials: Elena Roel Herranz, Principal Investigator — Public Health Agency of Barcelona
Locations (1):
- Agència de Salut Pública de Barcelona (ASPB), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] de Figueiredo A, Simas C, Karafillakis E, Paterson P, Larson HJ. Mapping global trends in vaccine confidence and investigating barriers to vaccine uptake: a large-scale retrospective temporal modelling study. Lancet. 2020 Sep 26;396(10255):898-908. doi: 10.1016/S0140-6736(20)31558-0. Epub 2020 Sep 10. PMID 32919524
- [Background] MacDonald NE; SAGE Working Group on Vaccine Hesitancy. Vaccine hesitancy: Definition, scope and determinants. Vaccine. 2015 Aug 14;33(34):4161-4. doi: 10.1016/j.vaccine.2015.04.036. Epub 2015 Apr 17. PMID 25896383
- [Background] Scalia P, Durand MA, Elwyn G. Shared decision-making interventions: An overview and a meta-analysis of their impact on vaccine uptake. J Intern Med. 2022 Apr;291(4):408-425. doi: 10.1111/joim.13405. Epub 2021 Nov 26. PMID 34700363
- [Background] Kok G, Gottlieb NH, Peters GJ, Mullen PD, Parcel GS, Ruiter RA, Fernandez ME, Markham C, Bartholomew LK. A taxonomy of behaviour change methods: an Intervention Mapping approach. Health Psychol Rev. 2016 Sep;10(3):297-312. doi: 10.1080/17437199.2015.1077155. Epub 2015 Oct 15. PMID 26262912
- [Background] Limaye RJ, Opel DJ, Dempsey A, Ellingson M, Spina C, Omer SB, Dudley MZ, Salmon DA, Leary SO. Communicating With Vaccine-Hesitant Parents: A Narrative Review. Acad Pediatr. 2021 May-Jun;21(4S):S24-S29. doi: 10.1016/j.acap.2021.01.018. PMID 33958087
- [Background] Opel DJ, Heritage J, Taylor JA, Mangione-Smith R, Salas HS, Devere V, Zhou C, Robinson JD. The architecture of provider-parent vaccine discussions at health supervision visits. Pediatrics. 2013 Dec;132(6):1037-46. doi: 10.1542/peds.2013-2037. Epub 2013 Nov 4. PMID 24190677
- [Background] Chamberlain AT, Limaye RJ, O'Leary ST, Frew PM, Brewer SE, Spina CI, Ellingson MK, Dudley MZ, Orenstein WA, Donnelly MA, Riley LE, Ault KA, Salmon DA, Omer SB. Development and acceptability of a video-based vaccine promotion tutorial for obstetric care providers. Vaccine. 2019 May 1;37(19):2532-2536. doi: 10.1016/j.vaccine.2019.03.005. Epub 2019 Apr 5. PMID 30962093
- [Background] Brewer NT. What Works to Increase Vaccination Uptake. Acad Pediatr. 2021 May-Jun;21(4S):S9-S16. doi: 10.1016/j.acap.2021.01.017. PMID 33958099
- [Background] Lip A, Pateman M, Fullerton MM, Chen HM, Bailey L, Houle S, Davidson S, Constantinescu C. Vaccine hesitancy educational tools for healthcare providers and trainees: A scoping review. Vaccine. 2023 Jan 4;41(1):23-35. doi: 10.1016/j.vaccine.2022.09.093. Epub 2022 Nov 24. PMID 36437208
- [Background] Jamison KC, Ahmed AH, Spoerner DA, Kinney D. Best shot: A motivational interviewing approach to address vaccine hesitancy in pediatric outpatient settings. J Pediatr Nurs. 2022 Nov-Dec;67:124-131. doi: 10.1016/j.pedn.2022.08.012. Epub 2022 Sep 13. PMID 36108393
- [Background] Gagneur A, Bergeron J, Gosselin V, Farrands A, Baron G. A complementary approach to the vaccination promotion continuum: An immunization-specific motivational-interview training for nurses. Vaccine. 2019 May 6;37(20):2748-2756. doi: 10.1016/j.vaccine.2019.03.076. Epub 2019 Apr 3. PMID 30954309
- [Background] Reno JE, Thomas J, Pyrzanowski J, Lockhart S, O'Leary ST, Campagna EJ, Dempsey AF. Examining strategies for improving healthcare providers' communication about adolescent HPV vaccination: evaluation of secondary outcomes in a randomized controlled trial. Hum Vaccin Immunother. 2019;15(7-8):1592-1598. doi: 10.1080/21645515.2018.1547607. Epub 2019 Jan 16. PMID 30433845
- [Background] Uthoff SAK, Zinkevich A, Franiel D, Below M, Splieth H, Iwen J, Biedermann M, Heinemeier D, Ansmann L. A complex intervention on vaccination uptake among older adults (>/= 60 years) in Germany - a study protocol with a mixed methods design. BMC Prim Care. 2023 Jul 15;24(1):148. doi: 10.1186/s12875-023-02101-w. PMID 37452283
- [Background] Jarrett C, Wilson R, O'Leary M, Eckersberger E, Larson HJ; SAGE Working Group on Vaccine Hesitancy. Strategies for addressing vaccine hesitancy - A systematic review. Vaccine. 2015 Aug 14;33(34):4180-90. doi: 10.1016/j.vaccine.2015.04.040. Epub 2015 Apr 18. PMID 25896377
- [Background] Opel DJ, Robinson JD, Spielvogle H, Spina C, Garrett K, Dempsey AF, Perreira C, Dickinson M, Zhou C, Pahud B, Taylor JA, O'Leary ST. 'Presumptively Initiating Vaccines and Optimizing Talk with Motivational Interviewing' (PIVOT with MI) trial: a protocol for a cluster randomised controlled trial of a clinician vaccine communication intervention. BMJ Open. 2020 Aug 11;10(8):e039299. doi: 10.1136/bmjopen-2020-039299. PMID 32784263
- [Background] Elizondo-Alzola U, G Carrasco M, Pinos L, Picchio CA, Rius C, Diez E. Vaccine hesitancy among paediatric nurses: Prevalence and associated factors. PLoS One. 2021 May 19;16(5):e0251735. doi: 10.1371/journal.pone.0251735. eCollection 2021. PMID 34010321
- [Background] Picchio CA, Carrasco MG, Sague-Vilavella M, Rius C. Knowledge, attitudes and beliefs about vaccination in primary healthcare workers involved in the administration of systematic childhood vaccines, Barcelona, 2016/17. Euro Surveill. 2019 Feb;24(6):1800117. doi: 10.2807/1560-7917.ES.2019.24.6.1800117. PMID 30755298
- [Derived] Roel E, Henderson E, Valmayor S, Porthe V, Asensio A, Ramirez-Morros A, Bruna X, Pasarin MI, Rius C, Diez E; CONFIVAC Research Group. Effectiveness of CONFIVAC, an intervention to enhance paediatric nurses and paediatricians skills to promote vaccination: A mixed-methods cluster randomized trial. Vaccine. 2025 Aug 30;62:127603. doi: 10.1016/j.vaccine.2025.127603. Epub 2025 Aug 15. PMID 40818260
- See also: Book: Qualitative Research & Evaluation Methods — https://us.sagepub.com/en-us/nam/qualitative-research-evaluation-methods/book232962
- See also: Book: Designing and Conducting Mixed Methods Research — https://books.google.es/books/about/Designing_and_Conducting_Mixed_Methods_R.html?id=eTwmDwAAQBAJ&redir_esc=y
- See also: BooK: Planning Health Promotion Programs: An Intervention Mapping Approach, 4th Edition — https://www.interventionmapping.com/